CLINICAL TRIAL: NCT00001007
Title: A Multicenter Phase I Trial To Evaluate the Safety and Pharmacokinetics of Intravenous and Oral Zidovudine in Infants With Perinatal Human Immunodeficiency Virus (HIV) Exposure
Brief Title: A Study of Zidovudine in Infants Exposed to the HIV Before or Soon After Birth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 049; FDA 9D
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2003-01

CONDITIONS: HIV Infections
Keywords: Pregnancy; Pregnancy Complications, Infectious; Infant, Newborn, Diseases; Infusions, Intravenous; Drug Evaluation; Administration, Oral; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious; Infant, Newborn, Diseases; Acquired Immunodeficiency Syndrome | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To determine if intravenous (IV) and oral zidovudine (AZT) can be safely given to children aged 1 day to 3 months who were born to mothers with an HIV infection. Also to determine the correct dose of AZT for young children. Of a total of 908 pediatric AIDS cases, 78 percent have acquired HIV infection from a mother with HIV infection or at high risk for acquisition of HIV, and the number of cases in children is expected to increase over the next several years. AZT therapy may be effective in altering the course of the disease and decreasing the high mortality in these children. It is also possible that early intervention with AZT may prevent the establishment of HIV contracted before, during, or just after birth.

DETAILED DESCRIPTION:
Of a total of 908 pediatric AIDS cases, 78 percent have acquired HIV infection from a mother with HIV infection or at high risk for acquisition of HIV, and the number of cases in children is expected to increase over the next several years. AZT therapy may be effective in altering the course of the disease and decreasing the high mortality in these children. It is also possible that early intervention with AZT may prevent the establishment of HIV contracted before, during, or just after birth.

The children entered in this study receive oral and IV AZT. The first 6 children receive 2 IV doses and 2 oral doses over a 2-week period, then 4 weeks of continuous oral dosing (4 doses per day). The remaining 12 children receive

1 IV dose and 1 oral dose followed by 6 weeks of oral AZT (4 doses per day) and a second IV dose at the end of the study. Each child is under the care of a specialist in pediatrics and has a physical examination and laboratory tests before starting AZT and 6 times while taking AZT to make sure the drug is not having a toxic effect on the child. A single cerebrospinal fluid (CSF) sample is taken from the last 12 children entering the study, so that the level of the AZT reaching the brain can be measured. The child returns to the hospital or clinic 4 weeks after the end of therapy to make sure that there are no delayed toxic effects.

ELIGIBILITY:
Inclusion Criteria

Infant gestation period must have been = or > 36 weeks and birthweight must = or > 2000 grams. Active infection must not be present at the time of entry into the study although an HIV culture or P24 serum antigen determination must be obtained prior to study entry. The child must have a life expectancy greater than 3 months. Parents or guardian must be available to give informed consent.

Prior Medication:

Allowed on a case-by-case basis:

* Some essential supportive therapies including antibiotics.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Any of the following laboratory findings within 2 weeks of study entry.
* A total bilirubin > 2 times age-adjusted upper limit of normal.
* Liver transaminase values > 3 x upper limit of normal.
* Serum creatinine > 1.5 x upper limit of normal.
* Total granulocyte count < 1500 cells/mm3.
* Hemoglobin < 10 g/dl or hemoglobinopathy.
* A urine toxicology screen positive for any drug or chemical.
* Infants must not have hemoglobinopathy or active infection at entry.

Prior Medication:

Excluded within 2 months of study entry:

* Antiretroviral agents.
* Excluded within 4 weeks of study entry:
* Immunomodulating agents including steroids, interferon, isoprinosine, and interleukin.
* Immunoglobulin.
* Excluded within 2 weeks of study entry:
* Any other experimental therapy, drugs which cause prolonged neutropenia or significant nephrotoxicity, or rifampin / rifampin derivatives.
* Some essential supportive therapies including antibiotics may have infrequent or transient effects. These drugs will be considered on a case-by-case basis.

Prior Treatment:

Excluded within 2 weeks of study entry:

* Red blood cells or whole blood transfusion.
* Excluded within 4 weeks of study entry:
* Lymphocyte transfusions for immune reconstitution.

Infants may not be entered into the study during the first 2 weeks of life if their mother received methadone therapy during the last trimester of her pregnancy or used any known illicit drug. A maternal urine toxicology screen may be optionally performed prior to entry of the child, and children whose mothers have a screen which is positive for any drugs or chemicals may not be enrolled within 2 weeks of the positive screen.

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18

CONTACTS AND LOCATIONS:
Overall Officials: Modlin J, Study Chair
Locations (6):
- United States (6):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Stanford Univ School of Medicine, Stanford, California
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Boston Med Ctr, Boston, Massachusetts
  - Duke Univ Med Ctr, Durham, North Carolina

REFERENCES:
- [Background] Vance E, Guzman J, Bitar M, Kazanjian P. Clarithromycin and zidovudine pharmacokinetic study. Int Conf AIDS. 1994 Aug 7-12;10(2):201 (abstract no PB0816)
- [Background] Vance E, Watson-Bitar M, Gustavson L, Kazanjian P. Pharmacokinetics of clarithromycin and zidovudine in patients with AIDS. Antimicrob Agents Chemother. 1995 Jun;39(6):1355-60. doi: 10.1128/AAC.39.6.1355. PMID 7574530
- [Background] Boucher FD, Modlin JF, Weller S, Ruff A, Mirochnick M, Pelton S, Wilfert C, McKinney R Jr, Crain MJ, Elkins MM, et al. Phase I evaluation of zidovudine administered to infants exposed at birth to the human immunodeficiency virus. J Pediatr. 1993 Jan;122(1):137-44. doi: 10.1016/s0022-3476(05)83507-3. PMID 8419601
- [Background] Collart L, Blaschke TF, Boucher F, Prober CG. Potential of population pharmacokinetics to reduce the frequency of blood sampling required for estimating kinetic parameters in neonates. Dev Pharmacol Ther. 1992;18(1-2):71-80. PMID 1483365
- [Background] Polis MA, Piscitelli SC, Vogel S, Witebsky FG, Conville PS, Petty B, Kovacs JA, Davey RT Jr, Walker RE, Falloon J, Metcalf JA, Craft C, Lane HC, Masur H. Clarithromycin lowers plasma zidovudine levels in persons with human immunodeficiency virus infection. Antimicrob Agents Chemother. 1997 Aug;41(8):1709-14. doi: 10.1128/AAC.41.8.1709. PMID 9257746
- [Background] Balis FM, Pizzo PA, Eddy J, Wilfert C, McKinney R, Scott G, Murphy RF, Jarosinski PF, Falloon J, Poplack DG. Pharmacokinetics of zidovudine administered intravenously and orally in children with human immunodeficiency virus infection. J Pediatr. 1989 May;114(5):880-4. doi: 10.1016/s0022-3476(89)80158-1. PMID 2715903